CLINICAL TRIAL: NCT04477759
Title: A Phase I Trial of MR-Guided Dose-Escalated Hypofractionated Adaptive Radiation Therapy and Immunotherapy in Primary Metastatic or Very Locally Advanced Patients With Head and Neck Cancer
Brief Title: Dose-Escalated Hypofractionated Adaptive Radiotherapy for Head and Neck Cancer
Acronym: DEHART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Musaddiq Awan, Principal Investigator, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038841; R21CA256144 (NIH)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Neoplasm
Keywords: Radiotherapy; Atezolizumab; Targeted Radiation Therapy; Head and Neck Cancer; Cancer; Magnetic Resonance Guided Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: This study will use a time-to-event continual reassessment method (TITE-CRM) for assigning subjects to the radiation therapy dosages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- 50 Gray (Gy) Radiation Therapy with Concurrent Atezolizumab (Experimental): 50 Gy of ionizing radiation therapy will be administered in 15 fractions.
  Interventions: Radiation: 50 Gy Radiation Therapy; Drug: Concurrent Atezolizumab
- 50 Gray (Gy) Radiation Therapy (Experimental): 50 Gy of ionizing radiation therapy will be administered in 15 fractions.
  Interventions: Radiation: 50 Gy Radiation Therapy; Drug: Adjuvant Atezolizumab
- 55 Gray (Gy) Radiation Therapy (Experimental): 55 Gy of ionizing radiation therapy will be administered in 15 fractions.
  Interventions: Radiation: 55 Gy Radiation Therapy; Drug: Adjuvant Atezolizumab
- 60 Gray (Gy) Radiation Therapy (Experimental): 60 Gy of ionizing radiation therapy will be administered in 15 fractions.
  Interventions: Radiation: 60 Gy Radiation Therapy; Drug: Adjuvant Atezolizumab

INTERVENTIONS:
Radiation: 50 Gy Radiation Therapy — Ionizing radiation
  Arms: 50 Gray (Gy) Radiation Therapy; 50 Gray (Gy) Radiation Therapy with Concurrent Atezolizumab
Radiation: 55 Gy Radiation Therapy — Ionizing radiation
  Arms: 55 Gray (Gy) Radiation Therapy
Radiation: 60 Gy Radiation Therapy — Ionizing radiation
  Arms: 60 Gray (Gy) Radiation Therapy
Drug: Concurrent Atezolizumab — Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 4 weeks following the initiation of radiation treatment up to 1 year from radiation fraction 1.
  Other Names: Tecentriq
  Arms: 50 Gray (Gy) Radiation Therapy with Concurrent Atezolizumab
Drug: Adjuvant Atezolizumab — Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
  Other Names: Tecentriq
  Arms: 50 Gray (Gy) Radiation Therapy; 55 Gray (Gy) Radiation Therapy; 60 Gray (Gy) Radiation Therapy

SUMMARY:
Locoregional failure remains the principal mode of mortality in head and neck squamous cell carcinoma (HNSCC) treated with conventional chemoradiation therapy. Magnetic resonance-guided radiation therapy (MRgRT) allows for adaptive radiation dose escalation based on tumor response and may improve therapeutic outcomes while limiting toxicities.

This protocol evaluates a novel framework for radiation delivery with concurrent atezolizumab in patients with advanced HNSCC. Dose-Escalated Hypofractionated Adaptive Radiotherapy (DEHART) modifies radiation dose using MRgRT by escalating radiation dose to residual tumor while deescalating radiation dose to areas of tumor regression.

DETAILED DESCRIPTION:
Locoregional failure remains the principal mode of mortality in head and neck squamous cell carcinoma (HNSCC) treated with conventional chemoradiation therapy. Radiation dose escalation with hypofractionation has shown unparalleled local control in other malignancies, such as non-small cell lung cancer, but has been limited in HNSCC due to toxicity concerns. Magnetic resonance-guided radiation therapy (MRgRT) allows for adaptive radiation dose escalation based on tumor response and may improve therapeutic outcomes while limiting toxicities.

This protocol evaluates a novel framework for radiation delivery using MRgRT with concurrent atezolizumab in patients with advanced HNSCC. Unlike conventional radiotherapy, Dose-Escalated Hypofractionated Adaptive Radiotherapy (DEHART) modifies radiation dose using MRgRT by adapting the radiation plan during the course of treatment, escalating radiation dose to residual tumor while deescalating radiation dose to areas of tumor regression. The hypothesis is that DEHART will safely deliver ablative radiation doses in 15 fractions over 3 weeks while limiting both toxicity and the effect of tumor repopulation by resistant clonogens, thus resulting in an improved therapeutic ratio.

This Phase I clinical trial will encompass the following specific aims: (1) determine the maximum tolerated dose (MTD) of the DEHART regimen delivered using MRgRT with concurrent atezolizumab in a population of patients who are not candidates or unsuitable for definitive chemoradiation therapy; (2) evaluate the toxicity and functional outcomes of the DEHART regimen; and (3) assess the efficacy of DEHART and obtain volumetric and functional imaging correlates of efficacy using MRgRT to serve as hypothesis-generating data for future trials of radiation dose adaptation. A modified Time-to Event Continual Reassessment (TITE-CRM) Phase I Design with three radiation dose levels delivered to regressing disease will be used to determine the MTD: 50 Gy in 15 fractions, 55 Gy in 15 fractions and 60 Gy in 15 fractions.

If DEHART is found to be safe and shows a signal of efficacy in this study, a future Phase II trial will be conducted to compare this novel treatment strategy to standard-of care conventionally fractionated chemoradiation in patients with locally advanced HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of T3-T4 N0-N3 M0 or T0-T4 N1-N3 M0 squamous cell carcinoma of the head and neck squamous cell carcinoma of the larynx, hypopharynx, oropharynx, oral cavity, or carcinoma of unknown head/neck primary) based on American Joint Committee on Cancer guideline (AJCC; 8th edition) with measurable disease who meet at least 1 one of the following 3 criteria:

  1. Not a candidates for concurrent, bolus, cisplatin-based chemoradiation therapy based on one of the following criteria (a-e)
  1. Age ≥ 70 with moderate to severe comorbidity or vulnerability to cisplatin, defined as having one or more of the following conditions within 4 week of registration:

     1. Modified Charlson Comorbidity Index ≥ 1
     2. Adult Comorbidity Evaluation-27 (ACE-27) Index ≥ 1
     3. ω score < 0.80
     4. Geriatric 8 (G-8) score ≤ 14
     5. Cancer and Aging Research Group (CARG) Toxicity Score ≥ 30%
     6. Cumulative Illness Rating Scale-Geriatric (CIRS-G) Score ≥ 4
  2. Age < 70 with severe comorbidity or vulnerability to cisplatin, defined as having two or more of the following conditions within 4 weeks prior to registration:

     1. Modified Charlson Comorbidity Index ≥ 1
     2. ACE-27 Index ≥ 1
     3. ω score < 0.80
     4. G-8 score ≤ 14
     5. CARG Toxicity Score ≥ 30%
     6. CIRS-G Score ≥ 4
  3. Creatinine clearance < 60 cc/min by the Cockroft-Gault formula
  4. Pre-existing peripheral neuropathy
  5. Clinical need for a hearing aid or 25+ decibel shift over 2 contiguous frequencies on a pre-treatment hearing test

     2. Patient refuses concurrent cisplatin-based chemoradiation therapy

     3. Patient has recurrent disease after definitive surgical resection
* Any patient 18 years or older with primary metastatic (AJCC 8th edition T1-T4 N0-N3 M1) squamous cell carcinoma of the head and neck
* Zubrod performance status 0-3
* Measurable primary and/or nodal tumor in the head and neck region at the time of radiotherapy
* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up.
* Ability to tolerate multiple MRIs
* Adequate hematologic function within 14 days prior to registration defined as follows: Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3, platelets ≥ 100,000 cells/mm^3, hemoglobin ≥ 9.0 g/dl, lymphocyte count ≥500/mL. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable).
* Adequate hepatic function within 14 days prior to registration defined as follows: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 times institutional upper limit of normal, serum bilirubin ≤ 1.5 x institutional upper limit of normal.
* For patients not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
* Negative HIV test at screening{, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/μL, and have an undetectable viral load}.
* Negative hepatitis B surface antigen (HBsAg) test at screening.
* Inclusion of Covid-19 positive patients will be based on standard institutional protocol.
* Female patients must meet one of the following:

  * Postmenopausal for at least one year before the screening visit, or
  * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), or
  * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agree to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 150 days after the last dose of study agent, AND o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, post ovulation methods] and withdrawal are not acceptable contraception methods).
* Male patients, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

  * Practice effective barrier contraception during the entire study period and through 150 calendar days after the last dose of study agent, OR
  * Must also adhere to the guidelines of any study-specific pregnancy prevention program, if applicable, OR o Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptom-thermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Prior invasive malignancy within the past 3 years (except for non-melanomatous skin cancer, and early stage treated prostate cancer);
* Life expectancy less than 12 months
* Performance status Zubrod >3
* Inability to encompass all gross disease in 19 cm superior to inferior planning target volume to be treated on the MR LINAC
* MRI-incompatible foreign body
* Claustrophobia precluding ability to tolerate multiple MRIs
* MRI-incompatible pacemaker or implantable cardioverter defibrillator (ICD) placement
* Patients with Cochlear implant
* Patients with prior radiation therapy to the head and neck Note: Prior external beam radiotherapy is excluded, but Iodine 131 is allowed.
* Prior systemic therapy, including cytotoxic chemotherapy, biologic/targeted therapy, or immune therapy for the study cancer
* Major surgery within 28 days prior to registration
* Body weight ≤ 30 kg
* Any of the following severe laboratory abnormalities within 14 days of registration, unless corrected prior to it: Sodium < 130 mmol/L or > 155 mmol/L; Potassium < 3.5 mmol/L or > 6 mmol/L ;Fasting glucose < 40 mg/dl or > 400 mg/dl;Serum calcium (ionized or adjusted for albumin) < 7 mg/dl or > 12.5 mg/dl; Magnesium < 0.9 mg/dl or > 3 mg/dl
* Unstable angina and/or congestive heart failure requiring hospitalization within 3 months prior to Step 1 registration
* Transmural myocardial infarction within 3 months prior to Step 1 registration
* Respiratory illness requiring hospitalization at the time of Step 1 registration
* Note: If the respiratory illness is resolved and the patient meets the eligibility status above, then the patient can be considered for the trial.
* Idiopathic pulmonary fibrosis or other severe interstitial lung disease that requires oxygen therapy or is thought to require oxygen therapy within 1 year prior to Step 1 registration
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Clinically apparent jaundice and/or known coagulation defects
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: Patients with vitiligo or alopecia; Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; Any chronic skin condition that does not require systemic therapy; Patients without active disease in the last 5 years may be included but only after consultation with the medical oncology study chair; Patients with celiac disease controlled by diet alone.
* History of active primary immunodeficiency including, but not limited to Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition. The need to exclude patients with AIDS from this protocol is necessary because the treatment involved in this protocol may be immunosuppressive. Patients with known HIV, cluster of differentiation 4 (CD4) cell counts ≥ 200/μL, and undetectable viral loads who are stable on an antiretroviral regimen may be included.
* Current or prior use of immunosuppressive medication within 14 days before registration, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Receipt of live attenuated vaccination within 30 days prior to registration
* Medical or psychiatric illness which would compromise the patient's ability to tolerate treatment or limit compliance with study requirements
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for 6 months after the last dose of atezolizumab, this exclusion is necessary because the treatment involved in this study may be significantly teratogenic. Women who are breastfeeding are also excluded.
* Prior allergic reaction or hypersensitivity to atezolizumab or any of study drug excipients.
* History of allogenic stem cell or organ transplantation
* Uncontrolled hypertension
* Uncontrolled cardiac arrhythmia
* Uncontrolled serious chronic gastrointestinal condition associated with diarrhea
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B viral (HBV) surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of leptomeningeal disease.
* Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurXâ) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia

  o Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Live, attenuated vaccines (e.g., FluMistâ) are prohibited within 4 weeks prior to initiation of study treatment, during treatment with atezolizumab, and for 5 months after the last dose of atezolizumab.
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, including anti-Cytotoxic T lymphocyte-associated antigen (anti-CTLA-4), anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 (IL-2) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the chemotherapy formulation
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Musaddiq Awan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab: 50 Gy of ionizing radiation therapy will be administered in 15 fractions. 50 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 4 weeks following the initiation of radiation treatment up to 1 year from radiation fraction 1.
- 50 Gray (Gy) Radiation Therapy With Adjuvant Atezolizumab: 50 Gy of ionizing radiation therapy will be administered in 15 fractions. 50 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
- 55 Gray (Gy) Radiation Therapy With Adjuvant Atezolizumab: 55 Gy of ionizing radiation therapy will be administered in 15 fractions. 55 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
- 60 Gray (Gy) Radiation Therapy With Adjuvant Atezolizumab: 60 Gy of ionizing radiation therapy will be administered in 15 fractions. 60 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
Period: Overall Study
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy With Adjuvant Atezolizumab | 55 Gray (Gy) Radiation Therapy With Adjuvant Atezolizumab | 60 Gray (Gy) Radiation Therapy With Adjuvant Atezolizumab
Started | 5 | 3 | 3 | 7
Completed | 5 | 3 | 3 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 50 Gray (Gy) Radiation Therapy: 50 Gy of ionizing radiation therapy will be administered in 15 fractions.
  50 Gy Radiation Therapy: Ionizing radiation
  Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 4 weeks following the initiation of radiation treatment up to 1 year from radiation fraction 1.
- 55 Gray (Gy) Radiation Therapy: 55 Gy of ionizing radiation therapy will be administered in 15 fractions.
  55 Gy Radiation Therapy: Ionizing radiation
  Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 4 weeks following the initiation of radiation treatment up to 1 year from radiation fraction 1.
- 60 Gray (Gy) Radiation Therapy: 60 Gy of ionizing radiation therapy will be administered in 15 fractions.
  60 Gy Radiation Therapy: Ionizing radiation
  Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 4 weeks following the initiation of radiation treatment up to 1 year from radiation fraction 1.
- Total: Total of all reporting groups
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy | 55 Gray (Gy) Radiation Therapy | 60 Gray (Gy) Radiation Therapy | Total
Number analyzed (Participants) | 5 | 3 | 3 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 1 | 6
  >=65 years | 4 | 1 | 1 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 3 | 7
  Male | 3 | 2 | 2 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 3 | 3 | 7 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 3 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-Limiting Toxicities at 50 Gy With Concurrent Atezolizumab
Description: This measure is the number of subjects experiencing a dose-limiting toxicity. A dose-limiting toxicity is defined as an inability to complete radiation treatment within 30 days of the start of radiotherapy that is not deemed to be related to disease progression; OR an unacceptable toxicity within one year of treatment (Grade 4+ toxicity) that is probably or definitely related to radiation treatment as determined by the treating physician or a death within one year of treatment that is probably or definitely related to treatment.
Time Frame: 12 months
Population: This applies only to this primary outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- 50 Gray (Gy) Radiation Therapy: 50 Gy of ionizing radiation therapy will be administered in 15 fractions. 50 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
- 55 Gray (Gy) Radiation Therapy: 55 Gy of ionizing radiation therapy will be administered in 15 fractions. 55 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
- 60 Gray (Gy) Radiation Therapy: 60 Gy of ionizing radiation therapy will be administered in 15 fractions. 60 Gy Radiation Therapy: Ionizing radiation Atezolizumab: Atezolizumab (1,680 mg) will be given to all subjects by intravenous injection every 28 days following the initiation of radiation treatment up to 1 year.
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy | 55 Gray (Gy) Radiation Therapy | 60 Gray (Gy) Radiation Therapy
Number analyzed (Participants) | 5 | 0 | 0 | 0
Participants | 2 | 0 | 0 | 0

2. Primary Outcome: Incidence of Dose-Limiting Toxicities at 50 Gy
Description: as for outcome 1
Time Frame: 12 months
Population: This applies only to this primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy | 55 Gray (Gy) Radiation Therapy | 60 Gray (Gy) Radiation Therapy
Number analyzed (Participants) | 0 | 3 | 0 | 0
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Dose-Limiting Toxicities at 55 Gy
Description: as for outcome 1
Time Frame: 12 months
Population: This applies only to this primary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy | 55 Gray (Gy) Radiation Therapy | 60 Gray (Gy) Radiation Therapy
Number analyzed (Participants) | 0 | 0 | 3 | 0
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Dose-Limiting Toxicities at 60 Gy
Description: as for outcome 1
Time Frame: 12 months
Population: This applies to this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy | 55 Gray (Gy) Radiation Therapy | 60 Gray (Gy) Radiation Therapy
Number analyzed (Participants) | 0 | 0 | 0 | 7
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Maximum Tolerated Radiation Dose
Description: This measure is the highest radiation dose at which there is a 30% or more rate of dose-limiting toxicity up to 12 months after completion of radiation treatment using the TITE-CRM design.
Time Frame: 12 months
Measure: Number; unit: Gy
Groups:
- All Participants: All participants who received a radiation dose either at 50 Gy, 55 Gy or 60 Gy.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Gy | 60

6. Secondary Outcome: Overall Survival
Description: This measure is the number of subjects alive at 1 year following the conclusion of scheduled radiation therapy.
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Locoregional Progression
Description: This measure is the number of subjects showing disease progression in the head and neck by RECIST criteria.
Time Frame: 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Gross Tumor Volume at Radiation Fraction 6 (Change From Baseline)
Description: This measure is the change in gross tumor volume for each subject as contoured on pre-treatment (baseline) and treatment 6 imaging scans. This will be measured in cubic centimeters.
Time Frame: 6th Radiation Fraction (approximately 1 week)
Reporting Status: Not Posted

9. Secondary Outcome: Gross Tumor Volume at Radiation Fraction 11 (Change From Baseline)
Description: This measure is the change in gross tumor volume for each subject as contoured on pre-treatment (baseline) and treatment 11 imaging scans. This will be measured in cubic centimeters.
Time Frame: 11th Radiation Fraction (approximately 2 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year following the end of radiation (up to 1 year and 3 weeks)
Description: regular investigator assessment, regular laboratory testing
Arm/Group | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab | 50 Gray (Gy) Radiation Therapy | 55 Gray (Gy) Radiation Therapy | 60 Gray (Gy) Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/3 | 1/3 | 2/7
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/3 | 2/3 | 6/7
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab (N=5) | 50 Gray (Gy) Radiation Therapy (N=3) | 55 Gray (Gy) Radiation Therapy (N=3) | 60 Gray (Gy) Radiation Therapy (N=7)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Hypercalcemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection - Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
arterial thromboembolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
G-tube malfunction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 Gray (Gy) Radiation Therapy With Concurrent Atezolizumab (N=5) | 50 Gray (Gy) Radiation Therapy (N=3) | 55 Gray (Gy) Radiation Therapy (N=3) | 60 Gray (Gy) Radiation Therapy (N=7)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (13) | 7 (15)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 7 (9)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (4) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 1 (2) | 5 (8)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 1 (1) | 2 (2) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (3) | 5 (7)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4)
Dysgeusia (Nervous system disorders) | 3 (4) | 3 (3) | 2 (4) | 4 (7)
Dysphagia (Gastrointestinal disorders) | 5 (11) | 3 (6) | 2 (3) | 7 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 1 (1) | 1 (3)
edema face (General disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (6) | 1 (4) | 3 (4) | 7 (10)
Fever (General disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thick secretions (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (5) | 1 (1)
Secretions (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
G-tube displacement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (6) | 4 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (9) | 0 (0) | 2 (4) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (5)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 5 (9) | 3 (8) | 3 (5) | 6 (15)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 4 (8) | 2 (3) | 1 (2) | 5 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck ococutaneous fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3) | 5 (7)
Thrush (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 5 (7)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 3 (4) | 1 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Weight loss (Investigations) | 3 (3) | 3 (7) | 1 (2) | 6 (16)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood tinged secretions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mouth swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mouth sore (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
G tube malfunction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
jaw pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Injury to carotid artery (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (10) | 6 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Transverse colon polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Open area anterior Right foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Left ear pain/pressure/popping (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucus/phlegm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cyst on left side of neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DVT in PICC line (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04477759/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04477759/ICF_001.pdf